CLINICAL TRIAL: NCT04761367
Title: Efficacy and Safety of PAIR Exercise Program After Total Hip and Knee Replacement: a Randomized Controlled Trial
Brief Title: Exercise Program After Total Hip and Knee Replacement: a Randomized Controlled Trial
Acronym: PAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1005/2020
Record Dates: First submitted 2021-02-05; First posted 2021-02-18 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Improve Quality of Life
Keywords: total knee replacement; total hip replacement; Physical activity; total knee prosthesis; total hip prosthesis
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION GROUP (Other): The IG will participate in a 6-month exercise program based on the PAIR exercise protocol and will receive educational sessions and material on the importance of maintaining an active life style after THR or TKR
  Interventions: Other: Physical activity. Physical Activity program is performed in a group in a gym
- CONTROL GROUP (No Intervention): The CG will receive only educational sessions and material on the importance of maintaining an active life style after THR or TKR

INTERVENTIONS:
Other: Physical activity. Physical Activity program is performed in a group in a gym — The intervention groups will be trained in a gyms under the direct supervision of a graduate trainer. All subjects will be requested to choose an additional third day of the week to carry out at least one of the following activities: walking, cycling or swimming
  Arms: INTERVENTION GROUP

SUMMARY:
Randomized controlled trial. Patients will be enrolled at the moment of the pre-surgery assessment after verifying the inclusion/exclusion criteria and signing written informed consent. After surgical treatment (THR or TKR) and subsequent rehabilitation treatment (which usually lasts 3-4 months) patients will be contacted and the persistence of inclusion/exclusion criteria verified again. For each type of surgical procedure (i.e. THR or TKR) those, with confirmed inclusion criteria will be randomly assigned to the IG or the CG. The IG will participate in a 6-month exercise program based on the PAIR exercise protocol and will receive educational sessions and material on the importance of maintaining an active life style after THR or TKR. The CG will receive only educational sessions and material on the importance of maintaining an active life style after THR or TKR. Participants of both IG and CG will be assessed at the moment of randomization (post-surgery baseline) and, subsequently, after 3 and 6 months.

DETAILED DESCRIPTION:
The present study is carried out within the project "Physical ActIvity after hip and knee Replacement" (PAIR) and funded within the Erasmus Plus Sport program (Grant Agreement 613008-EPP-1-2019-1-IT-SPO-SCP). It is aimed at evaluating the efficacy and safety of an exercise program specifically designed for improving physical function and QoL in people who had undergone THR or TKR for primary osteoarthritis after completing the surgical and rehabilitative treatment.

The primary objective of the study is to compare modifications of QoL measured with the Short-Form Health Survey (SF-36) induced in the intervention groups (IG) by the PAIR exercise program versus a control groups (CG) who will undergo usual care. SF-36 is one of the most widely used questionnaire to measure the health related QoL (HRQoL) in total hip and total knee arthroplasty patients.

The secondary objectives of the study are to investigate differences between IG and CG on domains which are considered to be determinants of QoL:

Hip- and knee-related impairments and functional limitations

* Harris Hip Score (HHS), American Knee Society scoring (KSS),
* Visual analog scale (VAS) to evaluate pain, High-Activity Arthroplasty Score (HAAS), ---Western Ontario and McMasters Universities Osteoarthritis
* Index (WOMAC),
* Knee Injury and Osteoarthritis Outcome Score (KOOS)
* Hip Disability and Osteoarthritis Score (HOOS).

Hip- and knee-related functional status

* Time Up and GO (TUG),
* Single Stance test,
* The 30-second Chair-Stand Test (30s-CST),
* Hand Grip test, Maximal strength of the lower limb,
* Hip and knee joints mobility (by goniometry).

Life style The ultimate goal of the PAIR exercise program is to increase physical activity in a sedentary population. The exercise program, through its beneficial effects on health, is expected to generate a virtuous circle promoting a more active life-style. For this domain 2 instruments will be used: Recent Physical Activity Questionnaire (RPAQ) and PAIR questionnaire for patients' attitudes toward physical (instrument generated within the PAIR project).

Safety: Adverse clinical events (ACEs) occurred to the participants both inside and outside gym classes.

Adherence: adherence of each subjects to the exercise program will be monitored in the IG. The adherence will be measured as percent of exercise sessions actually performed/total number of scheduled exercise sessions. Other factors considered to influence the adherence to an exercise program will be also recorded (age, gender, comorbidity, BMI, educational level, marital status, working activity, and home gym-distance).

Participants' satisfaction Satisfaction of PAIR exercise program is a very important domain since influence adherence. It will be verified by asking few questions with structured responses based on a 7-point Likert scale, to get participants' opinion about the PAIR exercise program.

ELIGIBILITY:
Inclusion Criteria:

Pre-surgery criteria

* Signed informed consent
* Age: 50-80 years
* Indications: Patient with unilateral advanced Osteo-Arthrosis (OA) requiring primary THR or TKR;
* General: American Society of Anesthesiologists (ASA) class 1 or 2
* Resident in Bologna metropolitan area

Post-surgery criteria

* Functional performance: Able to stand and walk >500 meters independently;
* Pain: score ≤ 4 in VAS

Exclusion Criteria:

* Unable/unwilling to sign the informed consent form of the study and/or willing to comply with the study requests
* Poor knowledge of Italian language which prevents understanding of the content of the consent form and/or of instructions for assessment and/or training;
* Severe functional limitations of other lower extremity joints besides that for which surgery is planned;
* Impairment of communicative and/or sensory functions so severe to make impossible understanding or executing trainer's instructions (dementia, aphasia, blindness, deafness);
* Heart failure (NYHA class >2);
* Unstable angina;
* Pulmonary disease requiring oxygen therapy;
* Symptomatic peripheral arteriopathy;
* Recent myocardial infarction or hospital admission for any other reason in the previous 6 months;
* Symptomatic orthostatic hypotension;
* Hypertension in poor pharmacologic control (diastolic >95 mmHg, systolic >160 mmHg);
* Relevant neurological condition impairing motor or cognitive function;
* Any other condition that the medical doctor (MD) considers to contraindicate the participation in an exercise program of moderate intensity;
* Severe depression.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaire | 6 months
  Short-Form Health Survey (SF-36). SF-36 is one of the most widely used questionnaire to measure the health related quality of life (QoL) items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100

SECONDARY OUTCOMES:
Clinical score about Hip | 6 months
  Harris Hip Score (HHS)41 is a disease-specific, health-related quality of life (HRQoL) instrument, widely used as an outcome measure after THR. The domains covered are pain, function, absence of deformity and range of movement
Clinical Score about Hip | 6 months
  American Knee Society scoring (KSS) is a disease-specific scoring system developed to assess clinical outcomes and functional ability on patients before and after total knee arthroplasty. Knees are examined for ROM, flexion contractures, extension leg, alignment and stability; functional score rates the patient's ability to walk and climb stairs.
Pain score | 6 months
  Visual analog scale (VAS) is scale to measure the pain
Lower limb function | 6 months
  High-Activity Arthroplasty Score (HAAS) focuses on lower limb functions and was specifically developed to assess the variations in functional ability after lower limb arthroplasty with particular regard to highly functioning individuals. The score is a 4-item self-assessment measure covering the 4 domains of walking, running, stair climbing, and general activities
Disability | 6 months
  Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC)47,48 is a valid and reliable scale, designed to provide a disease-specific measure for patients with osteoarthritis of hip and knee. It includes 24 items in three dimensions: pain (5 items), function (17 items) and stiffness (2 items).
Clinical outcome | 6 months
  Knee Injury and Osteoarthritis Outcome Score (KOOS) is a 42-item self-administered questionnaire which proved to be a reliable and valid instrument for evaluating the outcome of surgery and physical therapy50,51 for knee impairments. It includes subscales were sport and recreation function and knee-related QoL are considered. KOOS assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life.
Clinical score | 6 months
  Hip Disability and Osteoarthritis Score (HOOS),It is a 39-item self-administered questionnaire with five separate sub-scales: pain, symptoms, stiffness, activities of daily living, sport and recreation function, and hip-related quality of life
Physical performance | 6 months
  Time Up and GO (TUG) is a valid and reliable test used to examine physical performance and lower extremity
Balance | 6 months
  Single Stance test is useful to estimate standing balance and to discriminate from low to high functional ability in individuals of various ages and functional levels
Lower body strength | 6 months
  The 30-second Chair-Stand Test (30s-CST) is a valid and reliable single-item test for the assessment of lower body strength
Upper limb strength | 6 months
  Hand Grip test
Range of Motion (ROM) | 6 months
  Hip range of motion in degree, knee range of motion in degree, shoulder range of motion in degree

CONTACTS AND LOCATIONS:
Overall Officials: D Dallari, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No